CLINICAL TRIAL: NCT05325268
Title: Monteggia Fractures: Analysis of Patient Reported Outcome Measurements in Correlation to Ulnar Fracture Localization
Status: Completed | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Other Study IDs: Monteggia PROM
Record Dates: First submitted 2022-03-28; First posted 2022-04-13 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Monteggia's Fracture
Keywords: elbow; fracture; patient reported outcome
MeSH Terms: conditions — Monteggia's Fracture; Fractures, Bone | interventions — Fracture Fixation, Internal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Monteggia Cohort: Including all Patients. Patients who had suffered a Monteggia fracture and were treated with osteosynthesis
  Interventions: Procedure: Osteosynthesis

INTERVENTIONS:
Procedure: Osteosynthesis — Treatment of fracture with open reduction and osteosynthesis

SUMMARY:
Patients who had suffered a Monteggia fracture (lesion of the elbow) will be assessed regarding clinical and functional outcome (PROM) after treatment with osteosynthesis.

DETAILED DESCRIPTION:
A retrospective, monocentric study will be performed. Patients who underwent surgical treatment after suffering a Monteggia injury or a Monteggia like lesion between 2012 and 2018 will be included. Fractures will classified after Bado and Jupiter, according to the fracture location of the proximal ulna, as well as regarding the potential accompanying ligamentary injury.

In a follow-up examination validated patient-reported outcome measures (Disabilities of Arm, Shoulder and Hand Score [DASH], MEPS [Mayo Elbow Performance Score], Oxford Elbow Score [OES], Pain, Subjective Elbow Score) and functionality (range of motion [ROM], posterolateral instability, strength, valgus-/varus-stress) will be evaluated. In addition, treatment strategy and complications will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Monteggia fractures treated with osteosynthesis between 2012 and 2018
* understanding of German language (written and oral)
* informed consent

Exclusion Criteria:

* Patients not meeting the above criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated at the University Hospital Dresden.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Disabilities of Arm, Shoulder and Hand Score (DASH) | Time of Follow-Up assesment, approx. 3-7 years after surgery, avg. 50months
  Evaluation of the subjective function (patient reported outcome) using the DASH-Score, 0-100, best: 0, worst: 100
Oxford Elbow Score (OES) | Time of Follow-Up assesment, approx. 3-7 years after surgery, avg. 50months
  Evaluation of the subjective function (patient reported outcome) using the OES-Score, 0 - 48, best: 48, worst: 0
Mayo Elbow Performance Score (MEPS) | Time of Follow-Up assesment, approx. 3-7 years after surgery, avg. 50months
  Evaluation of the subjective function (patient reported outcome) using the MEPS-Score, 0-100, best: 100, worst: 0
Range of Motion (ROM) | Time of Follow-Up assesment, approx. 3-7 years after surgery, avg. 50months
  Objective functional clinical result. Evaluation of Motion of the Elbow in ° measured via goniometer. Physiological: Flexion/Extension 140/0/0°.

SECONDARY OUTCOMES:
Ulnar fracture localization (Radiologically) | baseline (timepoint of injury)
  Localization of ulnar fracture was measured from the proximal tip of the Olecranon to the fracture line on conventional X-ray in order to assess whether further distal fractures have a worse outcome compared to fractures with a close relation to or affecting the elbow joint [cm]

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinikum Carl Gustav Carus, Dresden, Germany

IPD SHARING:
Plan to Share IPD: No
No. Data may be shared upon reasonable request.

REFERENCES:
- [Derived] Tille E, Seidel L, Schlussler A, Beyer F, Kasten P, Bota O, Biewener A, Nowotny J. Monteggia fractures: analysis of patient-reported outcome measurements in correlation with ulnar fracture localization. J Orthop Surg Res. 2022 Jun 7;17(1):303. doi: 10.1186/s13018-022-03195-1. PMID 35672754